CLINICAL TRIAL: NCT02926794
Title: Reducing College Student Drinking by Integrating Self-Affirmation and Implementation Intentions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Santa Barbara (Other)
Responsible Party: Principal Investigator, Phillip Ehret, Graduate Student, University of California, Santa Barbara
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 38150394
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- SA and II (Experimental): Combined self-affirmation and implementations intention arm
  Interventions: Behavioral: SA and II
- SA and No II (Experimental): Self-affirmation and control intentions condition
  Interventions: Behavioral: SA and No II
- No SA and II (Experimental): Implementation intentions intervention and control writing task
  Interventions: Behavioral: No SA and II
- No SA and No II (Experimental): Control writing task and control intentions condition
  Interventions: Behavioral: No SA and No II

INTERVENTIONS:
Behavioral: SA and II — Self affirmation intervention where participants rank 11 values, then write about why their top ranked value is important AND Implementation intentions intervention where participants form two implementation intentions (If/then) statements regarding drinking behavior and write why these are important
  Arms: SA and II
Behavioral: SA and No II — Self affirmation intervention where participants rank 11 values, then write about why their top ranked value is important AND No implementation intentions intervention where participants write why selected health strategies are important (and do nothing else)
  Arms: SA and No II
Behavioral: No SA and II — Control writing intervention where participants rank 11 values, then write about why their 10th ranked value is important to someone else AND Implementation intentions intervention where participants form two implementation intentions (If/then) statements regarding drinking behavior and write why these are important
  Arms: No SA and II
Behavioral: No SA and No II — Control writing intervention where participants rank 11 values, then write about why their 10th ranked value is important to someone else AND No implementation intentions intervention where participants write why selected health strategies are important (and do nothing else)
  Arms: No SA and No II

SUMMARY:
Two hundred and ninety-three college students who reported drinking in the past month were randomly assigned to condition in a 2 (self-affirmation: values vs. control writing task) x 2 (implementation intentions: formed vs. not formed) between-subjects factorial design. Participants first completed a self-affirmation or control writing task, then read an article describing the risks of drinking. Next, all participants reported their common drinking behaviors and contexts, and then selected two harm-reduction strategies making either general intentions to use the strategies or making implementation intentions to use the strategies. Alcohol consumption was measured 1 and 2 weeks after the experimental session.

ELIGIBILITY:
Inclusion Criteria:

* Must have reported drinking at least 1 drink in the last 30 days at time of first participation.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | Past week drinking
  Number of standard drinks consumed in the past week

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ehret PJ, Sherman DK. Integrating Self-Affirmation and Implementation Intentions: Effects on College Student Drinking. Ann Behav Med. 2018 Jul 13;52(8):633-644. doi: 10.1093/abm/kax032. PMID 30010706